CLINICAL TRIAL: NCT01898858
Title: Effects of O2 and/or CO2 Inhalation on Rest and Exercise Pulmonary Hemodynamic
Acronym: H2PAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5546
Record Dates: First submitted 2013-06-21; First posted 2013-07-12 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Pulmonary Vascular Sensibility in Hypoxia; Hypercapnia; Hypoxia and Hypercapnia
MeSH Terms: conditions — Hypercapnia; Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HYPOXIA
  Interventions: Device: Hypoxia inhalation (Altitrainer NP 190)
- HYPERCAPNIA
  Interventions: Device: Hypercapnia inhalation (Altitrainer NP 190)
- HYPOXIA + HYPERCAPNIA
  Interventions: Device: Hypoxia and hypercapnia (Altitrainer NP 190)

INTERVENTIONS:
Device: Hypercapnia inhalation (Altitrainer NP 190) — Hypercapnia inhalation using an Altitrainer NP 190
  Groups: HYPERCAPNIA
Device: Hypoxia and hypercapnia (Altitrainer NP 190) — Hypoxia and hypercapnia inhalation using an Altitrainer NP 190
  Groups: HYPOXIA + HYPERCAPNIA
Device: Hypoxia inhalation (Altitrainer NP 190) — Hypoxia inhalation using an Altitrainer NP 190
  Groups: HYPOXIA

SUMMARY:
The aim of this study is to describe the pulmonary hemodynamic evolution at rest and during a short constant load exercise in 4 conditions :

* normoxia
* hypoxia
* hypercapnia
* association hypoxia and hypercapnia

ELIGIBILITY:
Inclusion criteria:

* healthy male
* exercise capacity between 100 and 130 % of theorical values

Exclusion criteria:

* smoker
* headache
* impossibility to perform an exercise test
* no tricuspid regurgitation on the echocardiography

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Systolic Artery Pulmonary Pressure(sPAP) (echocardiography, Cardiac output (impedancemetry), Cardiorespiratory parameters | at the end of the 30th minutes constant load exercise
  At rest and during exercise for each condition

SECONDARY OUTCOMES:
Dyspnea and muscle leg discomfort using a Borg Scale | at the end of the 30th minutes constant load exercise
  In each conditions at rest and during exercise

CONTACTS AND LOCATIONS:
Overall Officials: PISTEA Cristina, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Physiologie et d'Explorations Fonctionnelles, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg, France